CLINICAL TRIAL: NCT03465449
Title: Feasibility of Enhanced Dialysis Education (EDU) Intervention for Chronic Kidney Disease (CKD) Patients ≥ 75 Years of Age and Their Caregivers (CKD-EDU Study) - A Pilot Study
Brief Title: Feasibility of Enhanced Dialysis Education (EDU) Intervention for Chronic Kidney Disease (CKD) Patients
Acronym: CKD-EDU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Fahad Saeed, Assistant professor of medicine, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0071204
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual care (Active Comparator)
  Interventions: Other: usual care
- CKD-EDU arm (Experimental)
  Interventions: Behavioral: CKD-EDU

INTERVENTIONS:
Behavioral: CKD-EDU — Palliative Care based coaching intervention for support with dialysis-related decision making.
  Arms: CKD-EDU arm
Other: usual care — Nephrologist based usual care
  Arms: usual care

SUMMARY:
The investigators are studying the feasibility, acceptability, and outcomes of an intervention called Enhanced Dialysis Education (EDU) Intervention. CKD-EDU is a palliative care-based dialysis decision-making intervention that involves educating patients and caregivers about dialysis and engaging them in shared decision-making. Half of the enrolled patients will receive CKD-EDU and the other half will receive Usual Care.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥75 years old
2. Presence of advanced CKD stage 4 or 5 (i.e. e GFR ≤ 25 ml/min)
3. Patient's nephrologist is enrolled in the study and has seen that nephrologist at least once
4. Speaks English
5. Have not attended a dialysis education class or met with the dialysis education coordinator.
6. Have not made a dialysis decision

Exclusion Criteria:

1. Patient has already been seen by a palliative care clinician or is enrolled in hospice
2. Is already on dialysis
3. Hospitalized at the time of recruitment

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Number of participants receiving the intervention | 24 months
  We'll assess feasibility by determining the reach of the intervention
Acceptability of the intervention | 24 months
  We'll assess the acceptability of the CKD-PC intervention by qualitative interviews by reporting the percentage of patients with a favorable response to the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saeed F, Horowitz RK, Allen RJ, Auinger P, Epstein RM, Fiscella KA, Veazie PJ, Duberstein PR. Feasibility and Acceptability of a Palliative Care Intervention among Older Adults with Advanced CKD and Their Caregivers. Kidney360. 2025 Feb 1;6(2):236-246. doi: 10.34067/KID.0000000622. Epub 2024 Oct 24. PMID 40014547